CLINICAL TRIAL: NCT03615443
Title: Noninvasive vs. Invasive Lung Evaluation
Acronym: NILE
Status: Completed | Type: Observational
Sponsor: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GH03-001
Record Dates: First submitted 2018-07-13; First posted 2018-08-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment-naive metastatic non-squamous NSCLC
  Interventions: Diagnostic Test: Guardant360

INTERVENTIONS:
Diagnostic Test: Guardant360 — Guardant360 is a comprehensive, non-invasive tumor sequencing test.

SUMMARY:
Tumor derived cell free DNA (cfDNA) is increasingly used in the clinic to obtain genotype information about lung cancer, but its concordance with concurrent tumor-derived sequenced data is not known. The purpose of the trial is to determine the non-inferiority of cfDNA-based vs. tumor tissue-based genotyping as it pertains to the detection of National Comprehensive Cancer Network (NCCN)-recommended biomarkers in first line, treatment naive, non-squamous Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSCLC, which is: (1) Biopsy-proven (confirmatory biopsy must have been collected within 12 months prior to enrollment), (2) Metastatic (Stage IV, Stage IIIB when curative intent is not an option, or relapsed/recurrent disease after original diagnosis of Stage I-IIIA), (3) Non-squamous histology (mixed squamous and adenocarcinoma is allowed), (4) No prior treatment for advanced stage NSCLC: (a) Resection of or radiation to a single metastatic site is allowed if there are other untreated and measurable sites of metastatic disease at the time of enrollment. (b) Patients who have previously undergone surgical resection or radiation for Stage I-IIIA NSCLC are eligible if primary treatment was completed at least 6 months prior to the development of metastatic disease; for patients who received adjuvant systemic therapy, the last dose of treatment must be given at least 6 weeks prior to enrollment.
* Age ≥ 18 years
* Ability to understand a written informed consent document, and the willingness to sign it.
* Willingness to provide blood sample at the time points of pre-treatment, approximately 2 weeks after initiation of systemic treatment, and end of study).
* Patient has or will have standard-of-care tissue genotyping ordered. If the physician intends to order tissue genotyping, but there is insufficient material for analysis, the patient is still eligible for enrollment.

Exclusion Criteria:

* Pregnancy
* Any other concurrent malignancy except for localized, non-melanoma, cutaneous cancer or non-invasive cervical cancer. Any prior cancer other than NSCLC must have occurred more than 2 years prior to study entry with no evidence of currently active disease.
* Prior treatment for metastatic NSCLC including but not limited to: (1) Systemic treatment (targeted therapy, chemotherapy, immunotherapy, biologic therapy, etc.), (2) Resection of a metastatic lesion if the resected metastasis had been the only site of measurable metastatic disease, or resection of more than one metastatic lesion, (3) Radiation of a metastatic lesion or resection bed if given to the only measurable site of metastatic disease, or radiation to more than one metastatic lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve metastatic non-squamous non-small cell lung cancer (NSCLC).
Sampling Method: Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Demonstrate the non-inferiority of cfDNA-based vs. tumor tissue-based genotyping | 34 months
  The proportion of subjects for whom a genetic alteration is found in at least one of seven genes (EGFR, ALK, ROS1, BRAF, MET, ERBB2, RET) by testing tumor tissue will be compared to the proportion of subjects for whom a genetic alteration is found in at least one of the same genes by testing cfDNA.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 34 months
  The proportion of subjects with complete or partial tumor response as determined by the investigator. This will be assessed for the overall population and for the subpopulation of subjects who are identified by either tissue or cfDNA as having actionable EGFR activating mutations, ALK fusions, ROS1 fusions, and BRAF V600E mutations and who are subsequently treated with tyrosine kinase inhibitors.
Turnaround Time for cfDNA vs. Tissue Results | 34 months
  The time (in days) from the date of request for genetic testing to the report date for cfDNA and for tumor tissue.
Time to Treatment Initiation | 34 months
  The number of days from the date of study enrollment until the date that systemic or localized treatment is initiated.
Quantity Not Sufficient Rate of Tissue for Complete NCCN Biomarker Testing | 34 months
  The proportion of subjects deemed to have quantity not sufficient for tumor tissue testing of any of seven genes (EGFR, ALK, ROS1, BRAF, MET, ERBB2, RET) due to any of the following reasons: 1) insufficient tumor specimen for the genotyping tests to be performed, or 2) tumor cellularity below lab-dictated minimal requirements, or 3) no results available within 45 days of enrollment.
Tissue Incomplete Rate of Tissue for NCCN Biomarker Testing | 34 months
  The proportion of subjects with tumor tissue testing results not available for all seven genes (EGFR, ALK, ROS1, BRAF, MET, ERBB2, RET) and with no alterations detected among the genes that were tested.
Tumor Not Detected Rate of cfDNA in Blood | 34 months
  The proportion of subjects for whom cfDNA could not be detected in blood.
Sensitivity, Specificity, and Diagnostic Accuracy of Non-NCCN Biomarkers on the Guardant360 Panel | 34 months
  This objective applies to genes included in the Guardant360 panel other than EGFR, ALK, ROS1, BRAF, MET, ERBB2, RET and to subjects for whom both cfDNA and tumor tissue testing results are available. Diagnostic accuracy will include calculations for sensitivity, specificity, positive predictive value, and negative predictive value comparing tissue to cfDNA results and vice versa.
Rate of Discovery of Genomically Mediated, Acquired Resistance to Targeted Therapies in the Biomarker-Positive Subsets | 34 months
  Among subjects with tumor genetic alterations in EGFR, ALK, ROS1, BRAF, MET, ERBB2, or RET, the proportion with new (compared to baseline) genetic alterations in cfDNA at the time of disease progression following treatment with a therapy targeting the specific genetic alteration.

OTHER OUTCOMES:
Liquid Biopsy Rescue Rate of QNS Tissue Samples | 34 months
  Among subjects with tumor tissue quantity not sufficient for genetic testing, the proportion that had cfDNA detected.